CLINICAL TRIAL: NCT07341555
Title: IMMEDIATE EFFECTS OF SQUATS PERFORMED ON STABLE AND UNSTABLE SURFACES ON POSTURAL STABILITY, BILATERAL COMPARISON AND DYNAMIC BALANCE
Brief Title: Effect of Squats on Postural Stability, Bilateral Coordination and Dynamic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lithuanian Sports University28
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects
Keywords: postural balance; exercise; coordination
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group under three different conditions: no exercise, exercise on stable surface, and exercise on unstable surface.
Masking Description: No masking is applied in this study. This is a single-arm, open-label trial; therefore, no participants, care providers, investigators, or outcome assessors are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy student volunteers (Experimental): 42 students were tested under three conditions
  Interventions: Other: Condition - no exercise before testing; Other: Condition - exercise on unstable surface; Other: Condition - exercise on stable surface

INTERVENTIONS:
Other: Condition - no exercise before testing — Participants were tested without any exercise
Other: Condition - exercise on unstable surface — Participants performed 30 squats on unstable surface before testing
Other: Condition - exercise on stable surface — Participants performed 30 squats on stable surface before testing

SUMMARY:
The aim of this interventional study was to evaluate the immediate effects of a single bout of 30 squats performed on an unstable surface versus a stable surface on postural stability, bilateral coordination, and dynamic balance in healty subjects. We hypothesized that performing squats on an unstable surface would result in significantly greater improvements in these parameters compared to squats on a stable surface. By comparing the immediate effects under randomized conditions, this study seeks to contribute novel insights into the role of surface stability in acute exercise-induced balance adaptations.

DETAILED DESCRIPTION:
Despite the growing interest in instability training, there remains a lack of evidence regarding the acute effects of squats performed on stable versus unstable surfaces on key balance-related outcomes, including postural stability, bilateral coordination, and dynamic balance. Filling this gap is essential for informing clinical decision-making and optimizing performance and rehabilitation strategies. The study recruited young, relatively healthy, and physically active individuals-students (n = 42). Inclusion criteria were: 1) age between 18 and 35 years, and 2) voluntary consent to participate. Exclusion criteria were: 1) history of lower limb injury within the past six months, and 2) inability to maintain postural balance during testing.The study applied the following procedures: Participant Data Collection, Leg Length Measurement, Determination of Dominant Leg, Postural Stability Assesment, Dynamic Stability Assessment, and Bilateral coordination assessment.

All assessments were performed under controlled laboratory conditions by the same examiner to ensure reliability. Participants were instructed to avoid caffeine, strenuous exercise, and alcohol consumption for at least 12 hours prior to testing. and their hands placed on their hips.

Participants performed 30 bodyweight squats while standing with their feet shoulder-width apart and their hands placed on their hips. Each squat was executed to approximately 90° of knee flexion at the lowest point. The movements were paced using a metronome, with participants completing 30 squats within 45 seconds to ensure a consistent tempo and intensity.

The test was conducted under two conditions: on a stable surface and on an unstable surface, with a 48-hour interval between the two sessions.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 35 years,
2. voluntary consent to participate in the study.

Exclusion Criteria:

1. history of lower limb injury within the past six months,
2. inability to maintain postural balance during testing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Postural stability | Under three conditions (Condition 0, condition 1 an Condition 3) at least 48 hours apart
  Individuals were asked to stand on the platform with both feet barefoot; the platform's instabil-ity level was set to 11 (with 11 representing a predefined setting on the system). Foot position was determined using the Biodex Balance System (BBS) platform, with the cuboid bones serv-ing as anatomical landmarks to ensure that the foot was centred; subjects' arms were positioned on their hips throughout testing. Postural stability tests were measured in 10-second trials with a 10-second rest period between tests, with a total of three trials conducted.
  1. Stability index (the lower the index, the better the stability). Overall stability index (Overall), sagittal plane's stability index (Forward/Backward) and frontal plane's stability index (Left/Right).
  2. Sway index (the lower the index, the lower the sway)
  3. Time in Zone (four zone sizes in percentage provided).
  4. Time in Quadrant (percentage of time).
Bilteral Coordination | Under three conditions (Condition 0, condition 1 an Condition 3) at least 48 hours apart.
  Using the Biodex machine the following parameters were measured:
  1. Sway index in sagittal plane (Anterior/Posterior direction) while standing on a left leg, hand placed on hips. Lower index meant greater results.
  2. Sway index in sagittal plane (Anterior/Posterior direction) while standing on a right leg, hands placed on hips. Lower index meant greater results.
  3. Differences in the sway index in the sagittal plane between the two legs. Lower index meant greater results.
  4. Sway index in frontal plane (Medial/Lateral direction) while standing on a left leg, hands placed on hips. Lower index meant greater results.
  5. Sway index in frontal plane (Medial/Lateral direction) while standing on a right leg, hands placed on hips. Lower index meant greater results.
  6. Differences in the sway index in the frontal plane between the two legs. Lower index meant greater results.
  7. Overall sway index on the left leg.
  8. Overall sway index on the right leg.

SECONDARY OUTCOMES:
Dynamic balance | Under three conditions (Condition 0, condition 1 an Condition 3) at least 48 hours apart
  For Dynamic balance Y Balance test was used. Three attempts each leg were conducted, to anterior, poster-omedial and posterolateral directions. The mean of all three reaches were analysed. Participants were instructed to stand barefoot, maintain a single-leg stance and extend the contralateral leg to reach as far as possible along specified lines. The supporting leg could not move, hands were placed on the hips. Y Balance test's score was calculated using this formula: Normalized Reach Distance = (Sum of reach distances in three directions: Limb length) × 100.
Body hight | Befor testing
  in cm
Body weight | Before testing
  in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Department of health promotion and rehabilitation, Kaunas, Kauno M. Sav., Lithuania

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data, as the consent obtained from participants does not include permission for data sharing with other researchers.